CLINICAL TRIAL: NCT04840394
Title: Phase 1 Open-Label Dose Escalation Study of BDB001 as a Single Agent and in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Brief Title: Clinical Study of BDB018: Monotherapy and in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eikon Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BDB018-101; KEYNOTE-D26 (Other: Merck Sharp & Dohme Corp)
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Tumor, Solid
Keywords: TLR7/8; Immuno-oncology; TLR 7/8 Agonist; EIK1001
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BDB018 in Monotherapy (Experimental): A single subject will be enrolled at each dose level in the single agent arm.
  Then dosage escalation will follow a traditional 3+3 dose escalation design.
  Each successive group of patients will be enrolled at an incrementally higher dosage until the Maximum Tolerable Dose (MTD) or Recommended Phase 2 Dose (RP2D) of single agent BDB018 is reached.
  Interventions: Drug: BDB018
- BDB018 in Combination with Pembrolizumab (Experimental): In the combination arm of the study, a standard 3+3 dose escalation design will be utilized for all dose levels.
  When the MTD or RP2D of single agent BDB018 is reached, the first dose level cohort of the combination arm will begin. Once the MTD or RP2D in combination has been determined, approximately twenty additional subjects will be enrolled in the expansion phase of the study.
  Interventions: Drug: BDB018; Drug: Pembrolizumab

INTERVENTIONS:
Drug: BDB018 — BDB018 is an immunotherapy agent.
Drug: Pembrolizumab — Pembrolizumab is a potent humanized monoclonal antibody with high specificity of binding to the PD 1 receptor. Pembrolizumab has an acceptable preclinical safety profile and is approved as an IV therapy for a variety of advanced malignancies.
  Arms: BDB018 in Combination with Pembrolizumab

SUMMARY:
A Phase 1 Open-label Dose Escalation Trial of BDB018 in Monotherapy and in Combination with Pembrolizumab in Subjects with Advanced Solid Tumors

DETAILED DESCRIPTION:
This clinical trial is a study of an experimental drug called BDB018. BDB018 is a next-generation Toll-like receptor (TLR) 7/8 agonist that activates the immune system.

The primary objectives of this study are to evaluate the safety and tolerability of BDB018 in monotherapy and in combination with pembrolizumab (Keytruda) in subjects with unresectable or metastatic solid tumors that have relapsed or are refractory to standard treatment or for which there is no approved therapy.

This is a multi-center, open-label, dose escalation/dose expansion Phase 1 study of BDB018 in monotherapy and in combination with pembrolizumab.

The study will be conducted in two separate but independent parts: a dose escalation part with BDB018 in monotherapy and in combination with pembrolizumab and a dose expansion part of BDB018 in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed advanced or metastatic solid tumors that have disease progression after treatment with all available therapies for metastatic disease that are known to confer clinical benefit, or are intolerant to treatment, or refuse standard treatment. Note: there is no limit to the number of prior treatment regimens
2. Evidence of progressive disease (PD) within 3 months of signing the informed consent form.
3. Have measurable disease

Exclusion Criteria:

1. Has disease that is suitable for local therapy administered with curative intent.
2. Prior exposure to TLR7 agonists, TLR8 agonists, TLR 7/8 dual agonists, and TLR9 agonists.

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: incidence of adverse events and any dose limiting toxicity | Up to 30 months
  Safety and tolerability of BDB018 in monotherapy and in combination with pembrolizumab as measured by the incidence of adverse events and any dose limiting toxicity

SECONDARY OUTCOMES:
Determine Maximum Tolerated Dose | From first dose to 21 days after first dose for each patient (cycle 1)
  Determination of the maximum tolerated dose by assessing the frequency of BDB018 related and BDB018 and pembrolizumab-related adverse events using CTCAE version 5.0 to categorize adverse event severity
Radiographic Determination of Tumor Response after BDB018 Dosing | Every 63 days (3 cycles) up to 30 months after the first dose for each patient (each cycle is 21 days)
  Radiographic determination of tumor response in subjects dosed with BDB018 and BDB018 and pembrolizumab combination therapy using irRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Harry Raftopoulos, MD, Study Chair — Eikon Therapeutics
Locations (3):
- United States (3):
  - Florida Cancer Specialists, Sarasota, Florida
  - START MidWest, Grand Rapids, Michigan
  - START, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No